CLINICAL TRIAL: NCT04212923
Title: EHealth Based Self-management Intervention for Chronic Kidney Disease Care in China
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, nhchavannes, MD, PhD, Professor of Primary Care Medicine, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 201707040096
Record Dates: First submitted 2019-12-18; First posted 2019-12-30 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Chronic Kidney Diseases
Keywords: eHealth; self-management; chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Medical Dashboard based self-management intervention (Experimental): Chronic kidney disease patients in the intervention group will receive the usual care plus the tailored 'Medical Dashboard' based self-management intervention.
  Interventions: Behavioral: Medical Dashboard based self-management intervention
- Usual care services (No Intervention): Chronic kidney disease patients in the comparison group will receive usual care consisting of personalised in- and outpatient treatment based on symptoms experienced and disease severity, as outlined in the Kidney Disease Improving Global Outcomes (KDIGO).

INTERVENTIONS:
Behavioral: Medical Dashboard based self-management intervention — Before the start of the intervention, chronic kidney disease patients and care providers will receive a face-to-face training session on the use of Medical Dashboard. To avoid contamination, Medical Dashboard will only be made accessible for participants in the intervention group via a secure password-protected registration process.
  Arms: Medical Dashboard based self-management intervention

SUMMARY:
The purpose of this study is to develop an evidence-based tailored eHealth self-management intervention for patients with chronic kidney disease in China, and test the impact on implementation and effectiveness of interventions.

DETAILED DESCRIPTION:
Interventions that support disease self-management (further referred to as 'self-management interventions') can have a significant impact on the health and quality of life of patients suffering from chronic conditions in general and chronic kidney disease (CKD) patients in specific. In the last decade, the use of electronic health (eHealth) technology in self-management interventions has become more and more popular. EHealth-based self-management interventions have been shown to improve health-related outcomes, such as blood pressure (BP) control and medication adherence, and found to be feasible and acceptable for CKD patients and care professionals. Hence, the use of eHealth self-management interventions for CKD patients has become increasingly popular. Knowledge of the implementation and effectivity of such interventions in China and other developing countries is, however, still lacking. Researchers from the Leiden University Medical Center (LUMC) developed 'Medical Dashboard', an eHealth intervention to help support and involve CKD patients in their disease self-management. We aim to tailor the evidence-based Dutch intervention 'Medical Dashboard' to the Chinese context and evaluate its implementation process and effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients: (1) aged over 18 years old; (2) diagnosis of chronic kidney disease; (3) Chinese speaking.
* Health care providers who work in the Department of Nephrology

Exclusion Criteria:

* Individuals unable to participate due to physical or mental disabilities.
* Individuals unable to write or read.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change of chronic kidney disease self-management behavior using Chronic Kidney Disease Self-Management (CKD-SM) instrument from baseline to 3, 6 and 9 months after randomization | 0 month (baseline), 3 months after randomisation, 6 months after randomisation, 9 months after randomisation (endpoint)
  The Chronic Kidney Disease Self-Management (CKD-SM) instrument with 29 items uses a four-point likert scale ranging from 1 (never) to 4 (always) to measure subjects' self-management behavior. Possible scores range from 29 to 116 points, with higher scores indicating better self-management behavior

SECONDARY OUTCOMES:
Change of blood pressure from baseline to 3, 6 and 9 months after randomization | 0 month (baseline), 3 months after randomisation, 6 months after randomisation, 9 months after randomisation (endpoint)
  Change of blood pressure will be measured from baseline to 3, 6 and 9 months after randomization. The blood pressure will be measured in mmHg with systolic blood pressure and diastolic blood pressure
Change of body weight from baseline to 3, 6 and 9 months after randomization | 0 month (baseline), 3 months after randomization, 6 months after randomization, 9 months after randomization (endpoint)
  Change of body weight will be measured from baseline to 3, 6 and 9 months after randomization. The body weight will be measured in kilograms
Change of glomerular filtration rate from baseline to 3, 6 and 9 months after randomization | 0 month (baseline), 3 months after randomisation, 6 months after randomisation, 9 months after randomisation (endpoint)
  Glomerular filtration rate is a test used to check how well the kidneys are working. Change of glomerular filtration rate will be measured from baseline to 3, 6 and 9 months after randomization. The glomerular filtration rate will be measured in mL/min per 1.73 m2
Change of serum albumin from baseline to 3, 6 and 9 months after randomization | 0 month (baseline), 3 months after randomisation, 6 months after randomisation, 9 months after randomisation (endpoint)
  Change of serum albumin will be measured from baseline to 3, 6 and 9 months after randomization. The serum albumin will be measured in g/L
Change of serum creatinine from baseline to 3, 6 and 9 months after randomization | 0 month (baseline), 3 months after randomisation, 6 months after randomisation, 9 months after randomisation (endpoint)
  Change of serum creatinine will be measured from baseline to 3, 6 and 9 months after randomization. The serum creatinine will be measured in μmol/L
Change of number of complications patients have from baseline to 3, 6 and 9 months after randomization | 0 month (baseline), 3 months after randomisation, 6 months after randomisation, 9 months after randomisation (endpoint)
  Change of number of complications patients have will be measured from baseline to 3, 6 and 9 months after randomization
Change of chronic kidney disease self-efficacy using Chronic Kidney Disease Self-efficacy (CKD-SE) scale from baseline to 3, 6 and 9 months after randomization | 0 month (baseline), 3 months after randomisation, 6 months after randomisation, 9 months after randomisation (endpoint)
  The Chronic Kidney Disease Self-efficacy (CKD-SE) scale is a 25-item self-administered scale that measures subjects' confidence. Responses range from no confidence (0) to the highest degree of confidence (10). Possible scores range from 0 to 250 points, with higher scores indicating greater levels of confidence
Change of chronic kidney disease illness perception using Brief Illness Perception Questionnaire (BIPQ) from baseline to 9 months after randomization | 0 month (baseline), 9 months after randomisation (endpoint)
  The Brief Illness Perception Questionnaire (BIPQ) is a nine-item scale designed to rapidly assess the cognitive and emotional representations of illness. This scale consists of eight items related to illness perception. In addition, patients are asked to identify the three most important factors that they believe have caused their illness. All of the items except the causal question are rated using a 0 to 10 response scale. Higher scores indicate stronger perceptions along that dimension. The scores of items 3, 4, and 7 are calculated and expressed as reverse scores in this scale. Possible scores range from 0 to 80 points, with higher scores indicating a more threatening view of the illness
Change of chronic kidney disease anxiety and depression status using the Hospital Anxiety and Depression Scale (HADS) from baseline to 3, and 9 months after randomization | 0 month (baseline), 3 months after randomisation, 9 months after randomisation (endpoint)
  Hospital Anxiety and Depression Scale (HADS) is used to determine the levels of anxiety and depression that a person is experiencing. It is a fourteen item scale that generates ordinal data. Seven items measure symptoms of anxiety and seven items measure symptoms of depression . Each item is coded from 0 to 3. Possible scores range from 0 to 21 points for sub-scale on anxiety or depression, with higher scores indicating greater levels of burden of anxiety or depression
Change of chronic kidney disease quality of life using the Kidney Disease Quality of Life 36-item short-form survey (KDQOL-36) from baseline to 9 months after randomization | 0 month (baseline), 9 months after randomisation (endpoint)
  The Kidney Disease Quality of Life 36-item short-form survey (KDQOL-36) is used to evaluate the health-related quality of life. It has 36 items. Possible scores range from 0 to 100 points, with higher scores indicating better health-related quality of life
Hospital admission | 9 months after randomisation (endpoint)
  The time to first acute hospital admission with an exacerbation of chronic kidney disease or death due to chronic kidney disease within nine months after randomisation
Change of healthcare utilisation from 3 months after randomisation to 9 months after randomisation | 3 months after randomisation, 9 months after randomisation (endpoint)
  The change of healthcare utilisation will be measured by using the number of hospitalisations and emergency room visits, primary and secondary care visits of patients
Change of cost-benefit data from 3 months after randomisation to 9 months after randomisation | 3 months after randomisation, 9 months after randomisation (endpoint)
  The cost-benefit analysis will be measured by using medical cost (e.g., cost of treatment, hospitalization rates minored as monetary terms), all costs delivering the interventions (e.g., materials used in the interventions)
The proportion of chronic kidney disease patients and care professionals reached by the implementation of interventions | Throughout the 9-month trial
  The proportion of chronic kidney disease patients and care professionals eligible to use our intervention program, excluded, invited, and enrolled in the intervention
The number of implementation completion tasks completed | Throughout the 9-month trial
  The implementation completion tasks will be made as a checklist, and the number of implementations tasks finished will be checked
The number of chronic kidney disease patients' and care providers' use of the intervention | Throughout the 9-month trial
  The number of chronic kidney disease patients' and care providers' use of materials or system

CONTACTS AND LOCATIONS:
Overall Officials: Niels Chavannes, Principal Investigator — Leiden University Medical Center
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shen H, van der Kleij R, van der Boog PJM, Chavannes NH. Developing a Tailored eHealth Self-Management Intervention for Patients With Chronic Kidney Disease in China: Intervention Mapping Approach. JMIR Form Res. 2024 Jun 13;8:e48605. doi: 10.2196/48605. PMID 38869943
- [Derived] Shen H, van der Kleij R, van der Boog PJM, Song X, Wang W, Zhang T, Li Z, Lou X, Chavannes N. Development and evaluation of an eHealth self-management intervention for patients with chronic kidney disease in China: protocol for a mixed-method hybrid type 2 trial. BMC Nephrol. 2020 Nov 19;21(1):495. doi: 10.1186/s12882-020-02160-6. PMID 33213398